CLINICAL TRIAL: NCT03421808
Title: Randomized Controlled Trial of EEG/fMRI Controlled TMS For Treating Depression
Brief Title: EEG Synchronized TMS Trial for Depression
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00074695; R21MH106775-01 (NIH)
Record Dates: First submitted 2018-01-23; First posted 2018-02-05 (Actual); Results first posted 2025-08-14 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Depression
Keywords: TMS; transcranial magnetic stimulation; brain stimulation
MeSH Terms: conditions — Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: In a double blind, randomized (1:1) trial enrolling only at MUSC over three years in 60 treatment resistant depressed patients, we hypothesize that daily prefrontal rTMS over 4-6 weeks with the initial TMS pulse of each train synchronized to the subject's alpha phase (SYNC TMS), will result in improvement in depression, and that these improvements will be greater than the improvements seen using the same form of treatment but not with the initial pulse synchronized (NON-SYNC TMS).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All subjects will get EEGS and TMS, but in one group the TMS pulses are synchronized to the EEG, and in the other not. There is no way for the subject or treater or anyone to detect who is in which arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- SYNC TMS (Experimental): Patients will receive daily left prefrontal transcranial magnetic stimulation (TMS), 120% MT, 3000 pulses/session, for 30 sessions. They will have EEG and the TMS will be delivered at their individual alpha frequency (IAF) (8-12 Hz) and the first TMS pulse in each train of 40 pulses will be synchronized with the EEG so that the TMS pulse fires during the rising phase of the alpha rhythm.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- Non-Sync TMS (Active Comparator): Patients will receive daily left prefrontal transcranial Magnetic stimulation (TMS), 120% MT, 3000 pulses/session, for 30 sessions. They will have EEG and the TMS will be delivered at their individual alpha frequency (IAF) (8-12 Hz) and the first TMS pulse in each train of 40 pulses will NOT be synchronized with the EEG so that the TMS pulse fires during the rising phase of the alpha rhythm. This is the way conventional TMS is delivered now and is FDA approved.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — TMS

SUMMARY:
Daily prefrontal TMS for depression, as developed by the PI, involves delivering TMS pulses to the prefrontal cortex and not assessing what the actual EEG phase is of the person's brain. In cardiology, in order to stimulate the heart effectively, one has to know the rhythm and phase of the heartbeat in order to perform cardioversion. The investigators wonder if it is important to time the brain stimulation with the phase of the person's brain. The brain has definite rhythms, and cycles through being excited or resting. A common EEG rhythm is alpha frequency. Theoretically, the effect of the TMS pulse might be diminished if it was delivered when the brain was temporarily cycling into an off state.

In the r21 part of this grant, the investigators designed and constructed a combined TMS/EEG/fMRI system. With that equipment the investigators found that TMS pulses have different effects deeper in the brain as a function of the EEG alpha phase. Pulses delivered during a rising phase produce larger blood flow changes deeper in the brain than do pulses delivered during a falling phase.

In the R33 phase of the grant the investigators now take that idea into a small clinical trial in depression to test if synchronized pulses have a larger clinical effect than do non-synchronized pulses.

DETAILED DESCRIPTION:
The investigators have completed the first R21 phase of this combined two phase grant. Essentially, the investigators succeeded in creating for the first time on planet Earth a fully working combined and integrated TMS-fMRI-EEG system, and then used that in healthy controls to show that the secondary effect of the TMS pulse is greater when it is delivered to the cortex during the rising phase of the EEG alpha wave for that person. The group then also showed that they can monitor a subject with EEG and then predict and time a TMS pulse to be able to hit this time window.

The goal of the R33 phase of this R21/R33 grant is to test the hypothesis that synchronized stimulation has clinical implications; specifically that the increased rACC inhibition due to increased cortical activation of the DLPFC by synchronizing the TMS pulse application to an individual patient's alpha rhythm will have a significant effect on the anti-depressive treatment response rate for TMS, sufficient to justify a future, more extensive clinical trial.

In this study, the investigators will look first at the BOLD activity from the rACC as a measure of target engagement because there is a substantial literature suggesting that reductions in activity in the rACC are an integral part of the depression network and may predict eventual antidepressant effect. 1-5 Moreover, the investigators and others have shown that stimulation of the left DLPFC causes a reciprocal change in rACC. 6-9. The studies proposed for the R33 will randomize a cohort of 60 medication free depressed patients to standard TMS treatment (NON-SYNC) or timing optimized TMS treatment (SYNC). For the later cohort the investigators will use the results of the R21 phase to measure the optimum timing of the TMS pulses with respect to each individual's EEG rhythms to maximize inhibition of the rACC following TMS. This will be done at entry into the trial and after the therapy is complete. Both experimental and control group will undergo these measurements but they will only be used in the former group. To enable the 4 week (5 days/wk) TMS treatment plan to be able to use this individually determined timing, the investigators will integrate a second EEG system with our treatment TMS unit. The R33 specific aims are:

Specific Aim 1: Integrate a similar EEG system with our treatment TMS scanner with similar feedback circuitry as that in SA 3 in the R21.

Specific Aim 2: Carry out a 4 week trial (2 extra weeks for responders but not remitters) of anti-depressive therapy randomized between optimum timed TMS (SYNC) and standardized non-synchronous TMS (NON-SYNC) in a cohort of depressed patients to estimate the success rate of such an optimized treatment.

This study will provide the data needed for a go/no-go decision on a full clinical trial for this potential novel therapy.

Hypothesis: In a double blind, randomized (1:1) trial enrolling only at MUSC over three years in 60 treatment resistant depressed patients, we hypothesize that daily prefrontal rTMS over 4-6 weeks with the initial TMS pulse of each train synchronized to the subject's alpha phase (SYNC TMS), will result in improvement in depression, and that these improvements will be greater than the improvements seen using the same form of treatment but not with the initial pulse synchronized (NON-SYNC). As this work is a first ever use of this technology, the investigators wish to compare the antidepressant effects to standard therapy to see if synchronization boosts the clinical effect. A power analysis for this number of subjects exists but the investigators are really most interested in comparing the overall outcome between the two groups, and looking at response predictors. Thus it is not a formal efficacy or even inferiority trial, rather a comparative early phase trial.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of unipolar major depressive disorder, in a current major depressive episode, without psychotic features
2. Pretreatment Hamilton score ≥ 20
3. Age between 21 and 70 years
4. Fixed and stable antidepressant medications for 3 weeks prior and during the rTMS trial. Limit on benzodiazapenes to lorazepam (or equivalent) up to 3 mg every day
5. Moderate level of resistance to antidepressant treatment in the current episode, defined as failure of 1-4 adequate medication trials or intolerance to at least 3 trials, and duration of current episode ≤ 3 years
6. No history of schizophrenia, schizoaffective disorder, other [non mood disorder] psychosis, depression secondary to a medical condition, mental retardation, substance dependence or abuse within the past year (except nicotine), bipolar disorder, psychotic features in this or previous episodes, amnestic disorder, dementia or MMSE ≤24, delirium, obsessive compulsive disorder, post-traumatic stress disorder, panic disorder
7. No current Vagus Nerve Stimulation
8. No history of failing to respond to an adequate course of ECT in this or any episode, and no ECT within the past 3 months
9. No contraindication to MRI
10. No contraindication to rTMS (history of neurological disorder or seizure (except induced by ECT), increased intracranial pressure, brain surgery, or head trauma with loss of consciousness for >15 minutes, implanted electronic device, metal in the head, or pregnancy)
11. No history of autoimmune, endocrine, viral, or vascular disorder. No unstable cardiac disease, uncontrolled hypertension, or sleep apnea
12. No active suicidal intent or plan, or history of attempt within the past 12 months
13. Willing to provide informed consent

Exclusion Criteria:

1. To ensure that baseline levels of depression severity are stable at the time of study enrollment, patients will be dropped if they show > 30% improvement in the HRSD score from the time of initial intake (e.g., screening) to the baseline assessment.
2. Patients must have a recordable alpha frequency.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2024-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark S George, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina Brain Stimulation Division, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 34 were consented but subjects had to have a prestudy TMS/fMRI scan. Only 28 patients made it to actual randomization, and only 24 patients completed the trial. Data are presented on those who actually were randomized and had SYNC TMS or UNSYNC TMS.
Period: Overall Study
Arm/Group | SYNC TMS | Non-Sync TMS
Started | 15 | 13
Completed | 12 | 12
Not Completed | 3 | 1
Not completed — COVID related problems | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SYNC TMS | Non-Sync TMS | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (12.1) | 44 (12.4) | 43 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 11 | 10 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24
Depression illness duration (weeks) [Mean (Standard Deviation); unit: weeks] | 91 (79.3) | 60 (50.4) | 87 (60.1)

OUTCOME MEASURES:

1. Primary Outcome: Remission Rate
Description: Depression Remission, as defined by the Hamilton Rating Scale for Depression, 24 item, score less than 10. Range is 0 to 52. Higher scores mean more severe depression.
Time Frame: At the 4th week of treatment (or 6 weeks in those who continue to 6 weeks).
Measure: Count of Participants; unit: Participants
Arm/Group | SYNC TMS | Non-Sync TMS
Number analyzed (Participants) | 12 | 12
Participants | 2 | 3
Statistical Analysis 1: Comparison: SYNC TMS; For categorical clinical remission data we performed a chi-square test on the IIT and completer sample using Graph-Pad Prism; Test type: Superiority; p = 0.6, Chi-squared

2. Secondary Outcome: Number of Participants With EEG Phase Synchronization Frequency Changes
Description: EEG phase synchronization will be assessed by collecting real-time EEG, and then calculating whether the person's EEG frequency changed after the first few pulses in the train to where the EEG then matches the TMS pulses exactly and all TMS pulses are delivered at precisely the same time in the EEG cycle.
  We investigated the relationship between the maximum percentage phase angle (i.e., the histogram peak in the circular space of phases) and the HAMD changes across sessions. this maximum percentage was our first measure of the robustness of (defined as the corresponding phase of the post-stimulation ITPC value in circular space) across the 6 weeks of treatment.
Time Frame: assessed at each treatment session up to 6 weeks, week 6 reported
Population: We analyzed only completers as we needed the full 30 sessions of EEG for complete analysis. We measured the degree of phase entrainment, as measured by the inter-trial phase coherence (ITPC) across treatment sessions for SYNC and UNSYNC patients. We also measured the entrainment phase , defined as the corresponding phase in the circular space of post-stimulation ITPC value (i.e., the phase at which the first maximum ITPC after rTMS pulse train occurs).
Measure: Count of Participants; unit: Participants
Arm/Group | SYNC TMS | Non-Sync TMS
Number analyzed (Participants) | 12 | 12
Participants | 3 | 1

3. Secondary Outcome: EEG-TMS-fMRI Bold Changes in Cingulate Cortex
Description: EEG-TMS-fMRI Bold changes in cingulate cortex. We will measure the BOLD fMRI changes that are caused by a TMS pulse over the prefrontal cortex, and determine whether they increase more after 4 weeks of therapy.
Time Frame: At the 4th week of treatment (or 6 weeks in those who continue to 6 weeks).
Population: No participants were included in the analysis population for this outcome due to incomplete imaging data and lack of funding to perform analysis. Imaging data will not be analyzed at any point in the future. Although imaging data were collected for some participants, the data were incomplete and insufficient for analysis due to technical limitations and lack of funding to complete post-processing. Therefore, no participants were included in the analysis population for this outcome.
Arm/Group | SYNC TMS | Non-Sync TMS
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The full extent of the trial, June 2019 until February 2022. For each subject this covered the time of clinical participation and 6 month follow-up. More specifically, this was the time of clinical participation (up to 6 weeks) and 6 month follow-up, approximately 7.5 months,
Arm/Group | SYNC TMS | Non-Sync TMS
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/13
Other Adverse Events (participants affected / at risk) | 4/15 | 4/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SYNC TMS (N=15) | Non-Sync TMS (N=13)
Headache (Nervous system disorders) | 4 (19) | 4 (22) — Headache during or after treatment, blinded at the time of treatment.

LIMITATIONS AND CAVEATS:
Limitations are a small sample, using the intrinsic alpha frequency in each group, and the preferred synchronization was done before the trial and may have changed over time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-07): https://cdn.clinicaltrials.gov/large-docs/08/NCT03421808/Prot_SAP_000.pdf